CLINICAL TRIAL: NCT03145428
Title: Evaluation of Monocyte Volume Width Distribution (MDW) for Early Detection of Sepsis or Developing Sepsis on the UniCell DxH800 Hematology Analyzer
Brief Title: Evaluation of Monocyte Volume Distribution Width (MDW) for Early Detection of Sepsis
Acronym: MDW
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C03747
Record Dates: First submitted 2017-05-04; First posted 2017-05-09 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Sepsis; Severe Infection
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: CBC-Diff Monocyte volume width distribution (MDW) — MDW measurement used to detect sepsis. Results will not be used to manage patients

SUMMARY:
The measurement of monocyte volume width distribution (MDW) is intended for use with adult patients presenting to the emergency department (ED), where a CBC with Differential has been ordered, as an aid in the early detection of patients with or developing sepsis. The study will establish the clinical performance of MDW for detection of sepsis in the ED.

DETAILED DESCRIPTION:
A prospective multi-center study to establish the clinical utility of the measurement of monocyte volume width distribution, a cell population parameter of the CBC-Differential, on the Beckman Coulter Unicel DxH analyzers. The study will validate the cut-off for the early detection of sepsis in an adult emergency room population where the standard of care included a CBC with Differential and will evaluate the diagnostic performance of the parameter.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-89 years) presenting to ED
* All races & ethnicities
* CBC with Differential performed upon presentation
* Subjects with at least 12 hours of follow-up in ED (or in-patient if admitted)

Exclusion Criteria:

* Previously enrolled
* Subjects discharged <12 hours form ED presentation

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients with suspicion who present to ED and for whom CBC with Diff is performed upon ED presentation.
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Identification of sepsis vs. non-sepsis, including SIRS and infection (non-SIRS) by adjudication based on the 2001 SCCM sepsis definition (sepsis-2) | 12 hours after presentation to the ED
  Determination of the diagnostic accuracy, area under the receiver operating characteristic curve

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Crouser ED, Parrillo JE, Martin GS, Huang DT, Hausfater P, Grigorov I, Careaga D, Osborn T, Hasan M, Tejidor L. Monocyte distribution width enhances early sepsis detection in the emergency department beyond SIRS and qSOFA. J Intensive Care. 2020 May 5;8:33. doi: 10.1186/s40560-020-00446-3. eCollection 2020. PMID 32391157